CLINICAL TRIAL: NCT06210893
Title: Upwards Laryngeal Handshake Technique and Simple Palpation for Locating the Cricoid Cartilage : a Randomized Comparative Study
Brief Title: Upwards Laryngeal Handshake Technique and Simple Palpation for Locating the Cricoid Cartilage
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Professor, SMG-SNU Boramae Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2023-1
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Technique for Locating the Cricoid Cartilage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional simple palpation (Active Comparator): The cricoid cartilage is located with simple palpation.
  Interventions: Other: The cricoid cartilage is located.
- Upwards laryngeal handshake technique (Experimental): The cricoid cartilage is located with upwards laryngeal handshake technique.
  Interventions: Other: The cricoid cartilage is located.

INTERVENTIONS:
Other: The cricoid cartilage is located. — The cricoid cartilage is located.

SUMMARY:
This study aims to compare upwards laryngeal handshake technique and simple palpation for locating the cricoid cartilage.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing general anesthesia

Exclusion Criteria:

* History of neck surgery
* Anatomical anomaly or skin lesion in the neck
* History of gastroesophageal reflux disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-02-26 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Success rate for the correct identification of the cricoid cartilage | At 1 minute after induction of anesthesia
  Identification of the cricoid cartilage is evaluated using ultrasound.

SECONDARY OUTCOMES:
Distance from the cricoid cartilage center | At 1 minute after induction of anesthesia
  Distance from the cricoid cartilage center to the identification of the cricoid cartilage is assessed.